CLINICAL TRIAL: NCT00515866
Title: A Phase I, Open Label, Study of the Safety and Tolerability of KU-0059436 in Combination With Gemcitabine in the Treatment of Patients With Advanced Solid Tumours
Brief Title: Study to Assess the Safety & Tolerability of a PARP Inhibitor in Combination With Gemcitabine in Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KU36-29; D0810C00005
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Pancreatic Neoplasms
Keywords: Advanced pancreatic cancer; Poly (ADP ribose) polymerases; Advanced Solid Tumours
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — olaparib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Gemcitabine + KU-0059436
  Interventions: Drug: KU-0059436 (AZD2281)(PARP inhibitor); Drug: Gemcitabine

INTERVENTIONS:
Drug: KU-0059436 (AZD2281)(PARP inhibitor) — oral
  Other Names: Olaparib
Drug: Gemcitabine — intravenous injection
  Other Names: Gemzar®; Gemcitabine HCL

SUMMARY:
The purpose of this study is to identify a safe and tolerable dose of the drug KU-0059436 that can be given in combination with gemcitabine chemotherapy for the treatment of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of pancreas
* Locally advanced or metastatic unresectable disease

Exclusion Criteria:

* No prior anti cancer chemotherapy, radiotherapy (except palliative >4 weeks prior to entry, endocrine or immunotherapy or use of other investigational agents;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-08; Primary Completion 2011-10 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) or a tolerable and effective dose of KU 0059436 in combination with gemcitabine | assessed at each visit

SECONDARY OUTCOMES:
To identify the dose-limiting toxicity of the combination therapy | assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Burris III, MD, Principal Investigator — The Sarah Cannon Cancer Center; Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca
Locations (4):
- United States (2):
  - Research Site, New York, New York
  - Research Site, Nashville, Tennessee
- United Kingdom (2):
  - Research Site, London
  - Research Site, Oxford

REFERENCES:
- [Derived] Bendell J, O'Reilly EM, Middleton MR, Chau I, Hochster H, Fielding A, Burke W, Burris H 3rd. Phase I study of olaparib plus gemcitabine in patients with advanced solid tumours and comparison with gemcitabine alone in patients with locally advanced/metastatic pancreatic cancer. Ann Oncol. 2015 Apr;26(4):804-811. doi: 10.1093/annonc/mdu581. Epub 2015 Jan 7. PMID 25573533